CLINICAL TRIAL: NCT05041842
Title: Treatment With Tucatinib in Addition to Pertuzumab and Trastuzumab in Patients With HER2-positive Metastatic Breast Cancer After Local Therapy of Isolated Brain Progression
Brief Title: Treatment With Tucatinib in Patients With an Isolated Brain Progression of a Metastatic Breast Cancer
Acronym: InTTercePT
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Seagen Inc. (Industry); ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-BCG-2011; 2020-005735-79 (EudraCT Number)
Record Dates: First submitted 2021-09-03; First posted 2021-09-13 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Breast Cancer With a Isolated Brain Progression
MeSH Terms: interventions — tucatinib; pertuzumab; Trastuzumab; Biosimilar Pharmaceuticals

STUDY DESIGN:
Intervention Model Description: Patients treated with pertuzumab and trastuzumab for metastatic breast cancer who will develop an isolated brain relapse treated with local treatment will receive tucatinib in addition to pertuzumab and trastuzumab. Tucatinib will be taken orally 300 mg twice a day, pertuzumab (420 mg) and trastuzumab (6 mg/kg) will be taken every 3 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tucatinib plus systemic treatment with or without hormone therapy (Experimental): Addition of tucatinib to the systemic treatment (pertuzumab and trastuzumab) with or without hormone therapy.
  Interventions: Drug: Tucatinib; Drug: Pertuzumab; Drug: Trastuzumab; Drug: Hormone therapy; Drug: Pertuzumab/ Trastuzumab

INTERVENTIONS:
Drug: Tucatinib — 300 mg orally twice daily
Drug: Pertuzumab — Initial loading: 840 mg Maintenance: 420 mg, 3-weekly
  Other Names: Perjeta®
Drug: Trastuzumab — Intravenous formulation :
  Initial loading: 8 mg/kg Maintenance: 6 mg/kg, 3-weekly
  Subcutaneous formulation:
  600 mg (fixed dose regardless of patient's body weight), 3-weekly
  Other Names: Herceptin® or Biosimilar
Drug: Hormone therapy — Anastrozole (1 mg/day) or letrozole (2.5 mg/day) or fulvestrant (2x250 mg at day 1 and day 15 then every 4 weeks after the first injection)
Drug: Pertuzumab/ Trastuzumab — Initial loading:
  1200 mg Pertuzumab / 600 mg Trastuzumab (regardless of body weight)
  Maintenance:
  600 mg Pertuzumab / 600 mg Trastuzumab (regardless of body weight), 3-weekly
  Other Names: Phesgo®

SUMMARY:
The overall survival of patients with metastatic breast cancer has steadily improved over the past decades, mainly due to advances in systemic treatment. Despite these advances, the development of brain metastases remains a serious and devastating complication that decreases quality of life and increases morbidity and mortality. The HER2CLIMB randomized study demonstrated that adding the investigational drug tucatinib to the standard treatment trastuzumab and capecitabine improved both progression-free survival and overall survival in people diagnosed with human epidermal growth factor 2 (HER2)-positive metastatic breast cancer, previously treated with trastuzumab, pertuzumab, and T-DM1. In patients with brain metastases, the 1-year progression-free survival was 25% in the tucatinib group and 0% in the placebo group.

These results suggest that tucatinib may be a new standard treatment for HER2-positive metastatic disease.

The aim of the non-randomized phase II study, InTTercePT, is to evaluate the effectiveness of adding tucatinib to trastuzumab and pertuzumab in the event of cerebral progression, after the end of local treatment.

DETAILED DESCRIPTION:
The overall survival of patients with metastatic breast cancer has steadily improved over the past decades, mainly due to advances in systemic treatment. Despite these advances, the development of brain metastases remains a serious and devastating complication that decreases quality of life and increases morbidity and mortality. More than a third of patients with HER2-positive breast cancer develop brain metastases during the course of the disease. For patients with isolated brain progression, local treatment is recommended whenever possible (stereotaxic radiosurgery and / or surgery) as well as the continuation of systemic treatment previously initiated even if the evidence of a benefit is weak.

After local treatment these patients will have a higher risk of progression (cerebral and systemic). Therefore, the question of whether systemic treatment should be continued or changed remains an open question.

In a pooled analysis of two phase 1b studies, patients who continued systemic treatment with tucatinib (in combination with T-DM1 or with trastuzumab and capecitabine) after treatment directed to the central nervous system demonstrated a better prognosis than that of patients who stopped tucatinib.

The HER2CLIMB randomized study demonstrated that adding the investigational drug tucatinib to the standard treatment trastuzumab and capecitabine improved both progression-free survival and overall survival in people diagnosed with HER2-positive metastatic breast cancer, previously treated with trastuzumab, pertuzumab, and T-DM1. In patients with brain metastases, the 1-year progression-free survival was 25% in the tucatinib group and 0% in the placebo group.

These results suggest that tucatinib may be a new standard treatment for HER2-positive metastatic disease.

We anticipate that adding tucatinib to the trastuzumab / pertuzumab regimen will control brain metastases, prolong progression-free survival, and improve patient quality of life.

The aim of the non-randomized phase II study, InTTercePT, is to evaluate the effectiveness of adding tucatinib to trastuzumab and pertuzumab in the event of cerebral progression, after the end of local treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, Age ≥18;
2. Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0-1;
3. Histologically confirmed HER2 positive breast cancer, with HER2 positive defined by in situ hybridization (ISH), immunohistochemistry (IHC), or fluorescence in situ hybridization (FISH) methodology;
4. Documented isolated brain progression (defined as new or progressive brain metastases with stable or responding systemic disease) under pertuzumab and trastuzumab treatment (with or without taxane) for metastatic disease (There is no limit to the number and size of brain metastasis);
5. Complete local treatment of brain progression (Surgery and/or radiation therapy) should have been completed no more than 12 weeks before inclusion and there is no clinical indication for immediate re-treatment with local therapy in the opinion of the investigator;
6. Able to undergo MRI scanning of the brain;
7. Normal renal function: creatinine <1.5 x upper limit of normal (ULN);
8. Adequate liver function: total bilirubin ≤1.5 ULN (unless documented Gilbert's syndrome); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 ULN (≤5 ULN in the presence of liver metastases);
9. Normal hematological function: Absolute neutrophil count (ANC) ≥1.5 x 10⁹/L; platelets count ≥100 x 10⁹/L; and hemoglobin ≥9.0 g/dL;
10. Adequate cardiac functions, including:

    * 12 Lead electrocardiograms (ECG) with normal tracing or non-clinically significant changes that do not require medical intervention
    * QT/Corrected QT interval (QTcF) ≤470 msec for woman and ≤450 msec for men (mean of replicate values, correction per institutional standard) on the ECG at the screening visit and a normal kalemia
    * Left ventricular ejection fraction (LVEF) ≥50%
    * No history of Torsades de Pointes or other symptomatic QTc abnormality
11. Resolution of all acute toxic effects of prior anti-cancer therapy or surgical procedures to NCI CTCAE version 5.0 Grade 1 or to baseline (except alopecia or others toxicities not considered a safety risk for the patient at investigator's discretion);
12. Stable dose of steroids at the time of enrolment;
13. Women of childbearing potential must have a negative pregnancy test (blood or urine test) within 14 days prior to inclusion;
14. Woman of childbearing potential and male patients must agree to use adequate contraception for the duration of trial participation and up to 7 months after completing treatment/therapy (association of trastuzumab, pertuzumab +/- tucatinib). Hormonal contraceptives such as birth control pills, patches, implants, or injections are not allowed in patients who are hormone receptor positive;
15. Patient must have signed a written informed consent form prior to any trial specific procedures. When the patient is physically unable to give their written consent, a trusted person of their choice, independent from the investigator or the sponsor, can confirm in writing the patient's consent;
16. Patients affiliated to the social security system (or equivalent);
17. Patient must be willing and able to comply with the protocol for the duration of the trial including scheduled visits, treatment plan, laboratory tests, and examinations including follow-up.

Exclusion Criteria:

1. Radiologic extra-cranial progression under pertuzumab and trastuzumab treatment, at the time of enrolment. The systemic disease must be stable or responding at the time of enrolment;
2. Proven leptomeningeal disease;
3. Any progressive brain lesion between the brain local treatment completion and the enrolment;
4. Poorly controlled seizures (more than 1/week);
5. Clinically significant cardiopulmonary disease;
6. Used of a strong cytochrome P450 (CYP)2C8 inhibitor within 5 half-lives of the inhibitor, or use of a strong CYP3A4 or CYP2C8 inducer within 5 days prior to first dose of study treatment. Use of sensitive CYP3A substrates should be avoided one week before enrollment and during study treatment
7. Previous treatment with a tyrosine kinase inhibitor;
8. Carriers of Hepatitis B or Hepatitis C or have other known chronic liver disease;
9. Positive for human immunodeficiency virus (HIV);
10. Known prior severe hypersensitivity to tucatinib or compounds chemically or/and biologically similar or any component in its formulation;
11. History of any other cancer (except non-melanoma skin cancer or carcinoma in-situ of the cervix) unless the patient has been in remission and off all other cancer therapy for at least 3 years;
12. Pregnant women or women who are breast-feeding;
13. Inability to swallow tablets or significant gastrointestinal disease which would preclude the adequate oral absorption of medications;
14. Person deprived of their liberty or under protective custody or guardianship or unable to give informed consent;
15. Participation in another therapeutic trial within the 30 days prior to tucatinib treatment initiation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2021-12-17 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival | 6 months
  The progression-free survival is defined as the proportion of patients with an objective tumor progression by imaging, or death from any cause, whichever occurs first at 6 months from inclusion. Progression will be determined locally by the investigator through the use of Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) in case of lesions identified at baseline. For patients without any evidence of evidence at inclusion, the progression will be defined as an appearance of a new lesion (measurable or not measurable).

SECONDARY OUTCOMES:
Overall Survival | Throughout study completion, up to 18 months
  Overall Survival is defined as the time interval between the date of inclusion in the study and the date of death (all causes). Patients not known to have died at the time of analysis will be censored at the last recorded date on which the patient was known to be alive
Brain Progression-Free Survival | Throughout study completion, up to 18 months
  Brain Progression-Free Survival is defined as the time interval between the date of inclusion in the study and the date of documented progression of the brain metastases. Tumor progression will be evaluated according to RECIST v1.1, as determined by investigator assessment, or as the appearance of a lesion for patients in complete response (CR) at the brain level at the inclusion. Patients who have not progressed at the time of analysis will be censored at the time of the latest date of assessment from their last evaluable RECIST assessment.
Overall brain metastasis response | Throughout study completion, up to 18 months
  In patients who are not in CR at the brain level after local treatment: Overall brain metastasis response is defined as the best overall response of the brain metastases during the study. Brain metastases response will be evaluated according to RECIST v1.1, as determined by investigator assessment.
Incidence of treatment-emergent Adverse Events | Throughout study completion, up to 18 months
  Adverse Events will be graded according to National Cancer Institute-common terminology criteria for adverse events (NCI-CTCAE) v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Bachelot, MD, Principal Investigator — Centre Leon Berard; Anne-Claire Hardy-Bessard, MD, Principal Investigator — Centre Armoricain d'Oncologie
Locations (16):
- France (16):
  - Institut de Cancérologie de l'Ouest - Site Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Georges François Leclerc, Dijon
  - Clinique Victor Hugo, Le Mans
  - Centre Leon Berard, Lyon
  - Hôpital privé Jean Mermoz, Lyon
  - Institut du cancer de Montpellier, Montpellier
  - Centre Antoine Lacassagne, Nice
  - CARIO - Centre Armoricain Radiothérapie Imagerie Médicale et Oncologi, Plérin
  - Centre Hospitalier Annecy Genevois, Pringy
  - Institut Jean Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire de Tours, Tours
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared at an individual level. Those data will be part of the study database including all enrolled patients.